CLINICAL TRIAL: NCT03685591
Title: A PHASE 1 DOSE ESCALATION AND EXPANSION STUDY EVALUATING SAFETY, TOLERABILITY AND PHARMACOKINETICS OF PF 06952229 IN ADULT PATIENTS WITH ADVANCED SOLID TUMORS
Brief Title: PF-06952229 Treatment in Adult Patients With Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The decision to stop enrollment was due to strategic considerations and not due to any specific safety reasons or request from a regulatory authority.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: C3881001; C3881001 (Other: Alias Study Number)
Record Dates: First submitted 2018-09-20; First posted 2018-09-26 (Actual); Results first posted 2024-06-26 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Breast Neoplasms; Prostate Neoplasms; Neoplasms, Squamous Cell; Melanoma; Mesothelioma; Pancreatic Neoplasms; Colorectal Neoplasms; Carcinoma, Renal Cell; Liver Neoplasms
Keywords: efficacy; safety; pharmacokinetics; dose escalation; dose expansion; open-label; TGFb; transforming growth factor beta; breast cancer; prostate cancer; CRPC; metastatic; advanced; adenocarcinoma
MeSH Terms: conditions — Breast Neoplasms; Prostatic Neoplasms; Neoplasms, Squamous Cell; Melanoma; Mesothelioma; Pancreatic Neoplasms; Colorectal Neoplasms; Carcinoma, Renal Cell; Liver Neoplasms; Camurati-Engelmann Syndrome; Neoplasm Metastasis; Adenocarcinoma | interventions — enzalutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (15):
- Dose Level 1 (Part 1A) (Experimental): PF-06952229 at 20mg twice daily (BID)
  Interventions: Drug: PF-06952229
- Dose Level 2 (Part 1A) (Experimental): PF-06952229 at 40 mg BID
  Interventions: Drug: PF-06952229
- Dose Level 3 (Part 1A) (Experimental): PF-06952229 at 80 mg BID
  Interventions: Drug: PF-06952229
- Dose Level 4 (Part 1A) (Experimental): PF-06952229 at 150 mg BID
  Interventions: Drug: PF-06952229
- Dose Level 5 (Part 1A) (Experimental): PF-06952229 at 250 mg BID
  Interventions: Drug: PF-06952229
- Dose Level 6 (Part 1A) (Experimental): PF-06952229 at 375 mg BID
  Interventions: Drug: PF-06952229
- Dose Level 7 (Part 1A) (Experimental): PF-06952229 at 500 mg BID
  Interventions: Drug: PF-06952229
- Dose Level 8 (Part 1A) (Experimental): PF-06952229 at 625 mg BID
  Interventions: Drug: PF-06952229
- Dose Level 9 (Part 1A) (Experimental): PF-06952229 at 750 mg BID
  Interventions: Drug: PF-06952229
- Prostate Cancer Dose Level 1 (Part 1B) (Experimental): PF-06952229 at 375 mg BID in combination with enzalutamide
  Interventions: Drug: PF-06952229; Drug: Enzalutamide
- Prostate Cancer Dose Level 2 (Part 1B) (Experimental): PF-06952229 at 500 mg BID in combination with enzalutamide
  Interventions: Drug: PF-06952229; Drug: Enzalutamide
- Prostate Cancer Dose Level 3 (Part 1B) (Experimental): PF-06952229 at 625 mg BID in combination with enzalutamide
  Interventions: Drug: PF-06952229; Drug: Enzalutamide
- Prostate Cancer Dose Level 4 (Part 1B) (Experimental): PF-06952229 at 750 mg BID in combination with enzalutamide
  Interventions: Drug: PF-06952229; Drug: Enzalutamide
- Prostate Cancer (Part 2A) (Experimental): PF-06952229 at recommended Phase 2 Dose BID
  Interventions: Drug: PF-06952229
- Prostate Cancer (Part 2B) (Experimental): PF-06952229 at recommended phase 2 dose BID in combination with enzalutamide
  Interventions: Drug: PF-06952229; Drug: Enzalutamide

INTERVENTIONS:
Drug: PF-06952229 — Oral 7 days on / 7 days off - 28 day cycles (Part 1)
Drug: Enzalutamide — Prostate Cancer (Part 2). 160mg, capsules, orally, daily
  Arms: Prostate Cancer (Part 2B); Prostate Cancer Dose Level 1 (Part 1B); Prostate Cancer Dose Level 2 (Part 1B); Prostate Cancer Dose Level 3 (Part 1B); Prostate Cancer Dose Level 4 (Part 1B)

SUMMARY:
A Phase 1 dose escalation and expansion study evaluating safety, tolerability and pharmacokinetics of PF-06952229 in adult patients with advanced solid tumors.

DETAILED DESCRIPTION:
This is a Phase 1, open label, multi center, multiple dose, dose escalation and expansion, safety, tolerability, PK, and pharmacodynamics study of PF 06952229 in previously treated patients with advanced or metastatic cancers that may have high TGFbeta signatures and EMT expression.

The study includes Parts 1A and 1B, which are dose-escalation for monotherapy and combination therapy with enzalutamide, respectively, and Parts 2A and 2B, which are dose expansion for monotherapy and combination therapy with enzalutamide, respectively.

ELIGIBILITY:
Inclusion Criteria:

1. For Part 1A: Histological or cytological diagnosis of a solid tumor that is advanced/metastatic, patients are intolerant to standard treatment, resistant to standard therapy or for which no standard therapy is available for the following tumor types:

   Breast cancer; Prostate cancer (mCRPC testosterone less than 50 ng/dL); Squamous cell cancer of the head and neck; Melanoma; Mesothelioma; Pancreatic cancer; Colorectal cancer; Renal cell carcinoma; Hepatocellular cancer.
2. For Part 1B:

   * histological or cytological diagnosis of mCRPC 3 Part 2A and Part 2B:
   * Histologically or cytologically confirmed prostate adenocarcinoma metastatic disease.
   * Effective castration with serum testosterone levels 0.5 ng/mL (1.7 nmol/L).
   * Having received 3 or more cycles of prior docetaxel therapy (before or after abiraterone).
   * Having PD while receiving abiraterone acetate within 12 months of abiraterone treatment initiation.
   * Progressive disease (PD) by:

     1. Progression in measurable disease per RECIST 1.1 criteria. Patient with measurable disease must have at least 1 lesion that can be accurately measured in at least 1 dimension (longest diameter to be recorded). Each lesion must be at least 10 mm when measured by computed tomography (CT) (CT scan thickness no greater than 5 mm) or magnetic resonance imaging (MRI). Lymph nodes should be greater than or equal to 15 mm in short axis. As defined by PCWG2, if lymph node metastasis is the only evidence of metastasis, it must be greater than or equal to 20 mm in diameter when measured by spiral CT or MRI. Previously irradiated lesions, primary prostate lesion, and bone lesions will be considered non-measurable disease, or
     2. Appearance of 2 or more new bone lesions (PCWG2). They must be confirmed by other imaging modalities (CT; MRI) if ambiguous results, or
     3. Rising PSA defined (PCWG2) as at least 2 consecutive rises in PSA to be documented over a reference value (measure 1) taken at least 1 week apart. • Prior abiraterone acetate must be stopped at least 2 weeks before study treatment.

4. Patients must have recently obtained archival tumor tissue available for submission to the sponsor (except for Part 2A - monotherapy dose expansion). Patients enrolled in Part 1 and Part 2 should have access to their archival formalin-fixed paraffin-embedded material, collected within 6 months of screening, containing tumor that is of diagnostic quality and representative of their diagnosed malignancy or whenever possible, consent to undergo a biopsy during screening. The sponsor should be contacted if obtaining a new biopsy is not medically feasible for approval to enroll, prior to initiating screening activities.

5. Patients entering the study in the subgroup(s) requiring mandatory pre- and on treatment tumor biopsies in Part 2A and 2B must have a tumor amenable to biopsy and consent to these planned biopsy procedures. The sponsor should be contacted if obtaining a pre-treatment and on treatment biopsies is not medically feasible for approval to enroll, prior to initiating screening activities.

6. Age 18 years or older 7. Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) 0 or 1. 8. Adequate bone marrow function (see Appendix 3), including:

* Absolute Neutrophil Count (ANC) greater than or equal to 1,500/mm3;
* Platelets greater than or equal to 100,000/mm3;
* Hemoglobin greater than or equal to 9 g/dL. 9. Adequate renal function, including serum creatinine less than or equal to 1.5 x upper limit of normal (ULN) or estimated creatinine clearance greater than or equal to 60 mL/min as calculated using the method standard for the institution. In equivocal cases, a 24 hour urine collection test can be used to estimate the creatinine clearance more accurately. In Part 2: Serum creatinine of less than or equal to 3.0 x upper limit of normal.

  10. Adequate liver function, including:
* Total serum bilirubin less than or equal to 0.5 x ULN unless the patient has documented Gilbert syndrome;
* Aspartate and alanine aminotransferase (AST and ALT) less than or equal to 2.5 x ULN less than or equal to 5.0 x ULN if there is liver involvement by the tumor;
* Alkaline phosphatase less than or equal 2.5 x ULN less than or equal to 5 x ULN in case of bone metastasis).

  11. Serum phosphate within normal range (if abnormal, must be nonclinically significant per the Investigator and approval for patient inclusion after agreement from sponsor.

  12. Resolved acute effects of any prior therapy to baseline severity or CTCAE Grade 1 except for alopecia and those listed in the specific exclusion criteria.

  13. For Part 1A monotherapy dose escalation: serum pregnancy test (for females of childbearing potential) negative at screening.

  14. For Part 1A monotherapy dose escalation: female patients of nonchildbearing potential must meet at least 1 of the following criteria:
* Achieved postmenopausal status, defined as follows: cessation of regular menses for at least 12 consecutive months with no alternative pathological or physiological cause; and must have a serum follicle stimulating hormone level confirming the postmenopausal state;
* Have undergone a documented hysterectomy and/or bilateral oophorectomy;
* Have medically confirmed ovarian failure. All other female patients (including female patients with tubal ligations) are considered to be of childbearing potential.

  15. Evidence of a personally signed and dated informed consent document indicating that the patient has been informed of all pertinent aspects of the study.

  16. Willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other procedures.

Exclusion Criteria

Patients with any of the characteristics/conditions listed below will not be included in the study:

Any labs may be repeated for confirmation. Only the lab result requiring confirmation must be repeated, not the entire panel.

1. For Parts 1B current or prior treatment with enzalutamide within 24 days prior to first dose

   For 2A, and 2B:
   * Prior chemotherapy other than docetaxel for prostate cancer, except estramustine, adjuvant/neoadjuvant treatment completed more than 3 years ago;
   * Less than 28 days elapsed from prior treatment with chemotherapy, immunotherapy, radiotherapy, or surgery to the time of study enrollment.
2. Central Nervous System (CNS) metastases, carcinomatous meningitis, or leptomeningeal disease as indicated by baseline brain MRI (or CT with contrast if MRI is medically contraindicated), clinical symptoms, cerebral edema, and/or progressive growth. If contrast is medically contraindicated, a non-contrast CT scan may be performed.
3. Patients with a history of CNS metastases or cord compression.
4. Liver metastases at baseline as evidenced by CT scan or MRI that may be at risk for bleeding, such as those that are greater than 1 cm,
5. Patients with advanced/metastatic, symptomatic, visceral spread, that are at risk of life threatening complications in the short term (including patients with massive uncontrolled effusions [pleural, pericardial, peritoneal], pulmonary lymphangitis, and over 50% liver involvement). Note: Patients with indwelling catheter for drainage, or requirement for drainage no more frequently than monthly will be allowed.
6. Any other active malignancy within 3 years prior to study entry, except for adequately treated basal cell or squamous cell skin cancer, or carcinoma in situ.
7. Patients with a history of clinically significant tumor bleeding (except for bleeding in a post-operative setting), coagulopathy or arterio-venous malformations (AVM) or aneurysms in the CNS, liver, lung or other major organ of the body. Patients with known Osler-Weber-Rendu disease, Hemophilia A, Hemophilia B (Christmas Disease), Von Willibrand's Disease, Factor 13 deficiency and Factor 7 deficiency, antibodies to Factors 8 and 7, history of other bleeding diatheses and abnormal INR values.
8. Evidence of a tumor that compresses or invades major blood vessels or tumor cavitation that in the opinion of the investigator is likely to bleed.
9. Major surgery within 4 weeks prior to first dose.
10. Prior organ transplantation including heart and allogeneic stem cell transplantation.
11. Radiation therapy within 4 weeks prior to study entry. Note: Patients who have received radiotherapy must have recovered from any reversible side effects, such as nausea and vomiting.
12. Last anti cancer therapy including investigational drug(s) within 28 days (or 5 half-lives, whichever is shorter) prior to study entry excluding hormonal therapy.
13. Active and clinically significant bacterial, fungal, or viral infection, including known hepatitis B virus (HBV), known hepatitis C virus (HCV), known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS) related illness. In equivocal cases, with positive serology, those patients with a negative viral load are potentially eligible provided the other entry criteria are met. Note: Inclusion of patients with well controlled HIV, HBV or HCV can be discussed with sponsor on a case by case basis.

    • COVID-19/SARS-CoV2: Refer to Appendix 8 for further information.
14. Any of the following in the previous 6 months: myocardial infarction, congenital long QT syndrome, Torsades de pointes, arrhythmias (including sustained ventricular tachyarrhythmia and ventricular fibrillation), right bundle branch block and left anterior hemiblock (bifascicular block), unstable angina, coronary/peripheral artery bypass graft, symptomatic congestive heart failure (New York Heart Association class III or IV), cerebrovascular accident, transient ischemic attack, or symptomatic pulmonary embolism; deep venous thrombosis (DVT); arterial occlusive disease; ongoing cardiac dysrhythmias of National Cancer Institute (NCI) CTCAE Grade 2 or higher , atrial fibrillation of any grade that is uncontrolled, or QTcF interval greater than 470 msec at screening. Note: There is an exception where a cardiac rhythm device/pacemaker is fitted and results in QTcF greater than 470 msec.
15. Anticoagulation therapy with heparin, low molecular weight heparin, vitamin K antagonists, anti-platelet agents, or factor Xa inhibitors throughout the study and for at least 28 days post the last dose of study treatment. (If anticoagulation therapy is medically indicated on trial, patients should stop treatment with PF-06952229. For those requiring temporary anticoagulant therapy, resumption of PF-06952229 treatment may be permitted after discussion with the Sponsor. In any other case, study treatment should be permanently discontinued, and the patient should enter the follow-up portion of the trial.)
16. Moderate or severe heart valve function defect including moderate or severe valve stenosis or regurgitation.
17. Evidence or history of septal aneurysm, other heart aneurysm, or any aneurysm of the major vessels.
18. Grade 3 or higher cardiac troponin I at baseline.
19. Left ventricular ejection fraction (LVEF) of less than or equal to 50% or significant valvular regurgitation.
20. Hypertension that cannot be controlled by medications (greater than 150/90 mmHg despite optimal medical therapy) or requiring more than 2 medications for adequate control.
21. Clinically significant non healing or healing wounds.
22. For patients entering the combination with enzalutamide arm, history of seizures other than isolated febrile seizure in childhood.
23. Has a history of a cerebrovascular accident or transient ischemic attack less than 6 months ago.
24. Known or suspected hypersensitivity to active ingredient/excipients of PF 06952229 or enzalutamide.
25. Other acute or chronic medical or psychiatric condition, including recent (within the past year) or active suicidal ideation or behavior or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for entry into this study.
26. Investigator site staff members directly involved in the conduct of the study and their family members, site staff members otherwise supervised by the investigator, or patients who are Pfizer employees, including their family members, directly involved in the conduct of the study.
27. For Part 1A Monotherapy Dose Escalation: Pregnant female patients; breastfeeding female patients; fertile male patients and female patients of childbearing potential who are unwilling or unable to use 2 highly effective methods of contraception as outlined in this protocol for the duration of the study and for at least 28 days after the last dose of investigational product.
28. For Part 1B Combination Dose Escalation, Part 2A Monotherapy Expansion, and Part 2B Combination Dose Expansion: fertile male patients and female partners of childbearing potential who are unwilling or unable to use 2 highly effective methods of contraception as outlined in this protocol for the duration of the study and for at least 28 days after the last dose for monotherapy (Part 2A) or for at least 3 months after the last dose for combination therapy (Part 1B and Part 2B).
29. Inability to consume or absorb study drug, including but not limited to:

    • Active inflammatory gastrointestinal (GI) disease, known diverticular disease or previous gastric resection or lap band surgery. Impairment of gastro intestinal function or GI disease that may significantly alter the absorption of PF 06952229, such as history of GI surgery with may result in intestinal blind loops and patients with clinically significant gastroparesis, short bowel syndrome, unresolved nausea, vomiting, active inflammatory bowel disease or diarrhea of CTCAE Grade greater than 1.
30. Current use or anticipated need for food or drugs that are known strong and moderate CYP3A4/5 inhibitors, including their administration within 10 days or 5 half lives of the CYP3A4/5 inhibitor, whichever is longer, prior to first dose of investigational product.
31. Current use or anticipated need for drugs that are known strong and moderate CYP3A4/5 inducers, including their administration within 10 days or 5 half lives of the CYP3A4/5 inducer, whichever is longer, prior to the first dose of investigational product (See Section 5.7).
32. Have initiated bisphosphonates or approved receptor activator of nuclear factor kappa B ligand (RANK L) targeted agents (for example, denosumab) less than 14 days prior to study entry, unless there is agreement with the medical monitor.
33. Active, known suspect suspected autoimmune diseases including inflammatory bowel disease (including ulcerative colitis and Crohn's disease), rheumatoid arthritis, systemic progressive sclerosis, systemic lupus erythematosus (SLE), autoimmune vasculitis (eg, Wegener's Granulomatosis), CNS or motor neuropathy considered to be of autoimmune origin (eg, Gullian Barre Syndrome, Myasthenia Gravis, Multiple Sclerosis).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2018-10-04 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2022-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (15):
- United States (15):
  - HonorHealth, Scottsdale, Arizona
  - UCLA Dept of Medicine -Hematology/Oncology,Santa Monica, Santa Monica, California
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Mass General/ North Shore Center for Outpatient Care, Danvers, Massachusetts
  - Dana-Farber Cancer Institute - Chestnut Hill, Newton, Massachusetts
  - OU Medical Center Presbyterian Tower, Oklahoma City, Oklahoma
  - Stephenson Cancer Center, Oklahoma City, Oklahoma
  - Sarah Cannon Research Institute - Pharmacy, Nashville, Tennessee
  - Tennessee Oncology, PLLC, Nashville, Tennessee
  - The Sarah Cannon Research Institute / Tennessee Oncology, PLLC, Nashville, Tennessee
  - The Sarah Cannon Research Institute, Nashville, Tennessee
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - NEXT Oncology, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Yap TA, Choudhury AD, Hamilton E, Rosen LS, Stratton KL, Gordon MS, Schaer D, Liu L, Zhang L, Mittapalli RK, Zhong W, Soman N, Tolcher AW. PF-06952229, a selective TGF-beta-R1 inhibitor: preclinical development and a first-in-human, phase I, dose-escalation study in advanced solid tumors. ESMO Open. 2024 Sep;9(9):103653. doi: 10.1016/j.esmoop.2024.103653. Epub 2024 Aug 29. PMID 39214047
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C3881001

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 42 participants were enrolled in the Part 1A and all were treated. A total of 7 participants were enrolled in Part 1B and all were treated.
Groups:
- Part 1A: PF-06952229 20mg Monotherapy: PF-06952229 was administered at a dose of 20 mg orally twice daily (BID) for 7 days on, 7 days off for each Cycle (one cycle = 28 days).
- Part 1A: PF-06952229 40mg Monotherapy: PF-06952229 was administered at a dose of 40 mg orally BID for 7 days on, 7 days off for each Cycle (one cycle = 28 days).
- Part 1A: PF-06952229 80mg Monotherapy: PF-06952229 was administered at a dose of 80 mg orally BID for 7 days on, 7 days off for each Cycle (one cycle = 28 days).
- Part 1A: PF-06952229 150mg Monotherapy: PF-06952229 was administered at a dose of 150 mg orally BID for 7 days on, 7 days off for each Cycle (one cycle = 28 days).
- Part 1A: PF-06952229 250mg Monotherapy: PF-06952229 was administered at a dose of 250 mg orally BID for 7 days on, 7 days off for each Cycle (one cycle = 28 days).
- Part 1A: PF-06952229 375mg Monotherapy: PF-06952229 was administered at a dose of 375 mg orally BID for 7 days on, 7 days off for each Cycle (one cycle = 28 days).
- Part 1A: PF-06952229 500mg Monotherapy: PF-06952229 was administered at a dose of 500 mg orally BID for 7 days on, 7 days off for each Cycle (one cycle = 28 days).
- Part 1B: PF-06952229 250mg + Enzalutamide: PF-06952229 was administered at a dose of 250 mg orally twice daily (BID) for 7 days on, 7 days off for each Cycle (one cycle = 28 days) in combination with enzalutamide at 160 mg orally once a day (QD) as continuous daily dosing.
- Part 1B: PF-06952229 375mg + Enzalutamide: PF-06952229 was administered at a dose of 375 mg orally twice daily (BID) for 7 days on, 7 days off for each Cycle (one cycle = 28 days) in combination with enzalutamide at 160 mg orally QD as continuous daily dosing.
Period: Overall Study
Arm/Group | Part 1A: PF-06952229 20mg Monotherapy | Part 1A: PF-06952229 40mg Monotherapy | Part 1A: PF-06952229 80mg Monotherapy | Part 1A: PF-06952229 150mg Monotherapy | Part 1A: PF-06952229 250mg Monotherapy | Part 1A: PF-06952229 375mg Monotherapy | Part 1A: PF-06952229 500mg Monotherapy | Part 1B: PF-06952229 250mg + Enzalutamide | Part 1B: PF-06952229 375mg + Enzalutamide
Started | 1 | 1 | 1 | 5 | 13 | 17 | 4 | 4 | 3
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 1 | 1 | 1 | 5 | 13 | 17 | 4 | 4 | 3
Not completed — Global Deterioration of Health Status | 0 | 0 | 0 | 1 | 2 | 4 | 1 | 1 | 0
Not completed — Progressive Disease | 1 | 1 | 0 | 3 | 5 | 4 | 3 | 2 | 1
Not completed — Other | 0 | 0 | 1 | 0 | 2 | 3 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 3 | 2 | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 1 | 4 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: All enrolled participants who received at least one dose of study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1A: PF-06952229 20mg Monotherapy | Part 1A: PF-06952229 40mg Monotherapy | Part 1A: PF-06952229 80mg Monotherapy | Part 1A: PF-06952229 150mg Monotherapy | Part 1A: PF-06952229 250mg Monotherapy | Part 1A: PF-06952229 375mg Monotherapy | Part 1A: PF-06952229 500mg Monotherapy | Part 1B: PF-06952229 250mg + Enzalutamide | Part 1B: PF-06952229 375mg + Enzalutamide | Total
Number analyzed (Participants) | 1 | 1 | 1 | 5 | 13 | 17 | 4 | 4 | 3 | 49
Age, Continuous [Median (Full Range); unit: Years] | 79.00 [79 to 79] | 74.00 [74 to 74] | 73.00 [73 to 73] | 65.00 [53 to 75] | 69.00 [26 to 76] | 67.00 [54 to 88] | 75.50 [72 to 78] | 61.50 [57 to 71] | 69.00 [58 to 69] | 69.00 [26 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 1 | 3 | 1 | 0 | 0 | 0 | 5
  Male | 1 | 1 | 1 | 4 | 10 | 16 | 4 | 4 | 3 | 44
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 3
  Not Hispanic or Latino | 1 | 1 | 1 | 4 | 10 | 14 | 4 | 4 | 3 | 42
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 1 | 1 | 1 | 4 | 11 | 14 | 3 | 3 | 2 | 40
  Black or African American | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 4
  Asian | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 2
  Not reported | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With First-Cycle Dose-Limiting Toxicitys (DLTs) by Treatment
Description: First cycle DLTs were utilized to determine the max tolerated dose and future escalations or deescalations. Any of the following adverse events occurred in the first cycle of treatment which were clinically significant were classified as DLTs: Hematologic: Thrombocytopenia Grade 4 for >=7 days, or Grade 3 or 4 associated with >= Grade 2 clinically significant bleeding or requiring platelet transfusion; Neutropenia Grade 4 for >=7 days; Grade>=3 neutropenia with infection; Anemia Grade 4 or Grade 3 requiring blood transfusion. Nonhematologic: Grade>=3 toxicities that were considered clinically significant; Alanine aminotransferase/aspartate aminotransferase>3x the upper limit of normal (ULN) with bilirubin>2x ULN without another explanation; Grade 3 nausea, vomiting or diarrhea that did not resolve within 4 days despite maximal supportive therapy. Nonhematologic and Non-Hepatic: Any toxicity caused>= 2 weeks of dose delay or preventing participants from receiving 75% of study drug.
Time Frame: Within 28 days of first dose or until the participant completed the first cycle of therapy if there were treatment delayed (on average 28 days).
Population: Population included all enrolled participants who received at least one dose of investigational product and included data evaluated for a minimum DLT observation period of 28 days.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1A: PF-06952229 20mg Monotherapy | Part 1A: PF-06952229 40mg Monotherapy | Part 1A: PF-06952229 80mg Monotherapy | Part 1A: PF-06952229 150mg Monotherapy | Part 1A: PF-06952229 250mg Monotherapy | Part 1A: PF-06952229 375mg Monotherapy | Part 1A: PF-06952229 500mg Monotherapy | Part 1B: PF-06952229 250mg + Enzalutamide | Part 1B: PF-06952229 375mg + Enzalutamide
Number analyzed (Participants) | 1 | 1 | 1 | 4 | 9 | 15 | 4 | 4 | 3
Participants | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0

2. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (Treatment Related)
Description: Treatment-related AE was any untoward medical occurrence attributed to study drug in a participant who received study drug. An SAE was an AE resulting in any of death; inpatient hospitalization; life-threatening experience; disability; congenital anomaly or deemed significant for any other reason. Symptoms of infusion-related reactions (IRRs) may include, but were not limited to, fever, chills, flushing, hypotension, dyspnea, wheezing, back pain, abdominal pain, and urticaria. Grade 3: severe or medically significant but not immediately life-threatening, hospitalization or prolongation of existing hospitalization indicated, disabling, limiting self-care ADL; Grade 4: life-threatening consequence, urgent intervention indicated; Grade 5: death related to AE.
Time Frame: Baseline up to 28 days after last dose of study treatment ( up to approximately 2 years)
Population: Population included all enrolled participants who received at least one dose of investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1A: PF-06952229 20mg Monotherapy | Part 1A: PF-06952229 40mg Monotherapy | Part 1A: PF-06952229 80mg Monotherapy | Part 1A: PF-06952229 150mg Monotherapy | Part 1A: PF-06952229 250mg Monotherapy | Part 1A: PF-06952229 375mg Monotherapy | Part 1A: PF-06952229 500mg Monotherapy | Part 1B: PF-06952229 250mg + Enzalutamide | Part 1B: PF-06952229 375mg + Enzalutamide
Number analyzed (Participants) | 1 | 1 | 1 | 5 | 13 | 17 | 4 | 4 | 3
Participants
  Participants with adverse events | 1 | 1 | 1 | 1 | 9 | 13 | 4 | 1 | 1
  Participants with serious adverse events | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 0
  Participants with Maximum Grade 3 or 4 adverse events | 0 | 0 | 0 | 1 | 2 | 6 | 3 | 1 | 0
  Participants with Maximum Grade 5 adverse events | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Participants discontinued from study due to adverse events | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 1 | 1
  Participants discontinued study drug due to AE and continue Study | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Participants with dose reduced or temporary discontinuation due to adverse events | 0 | 0 | 0 | 0 | 3 | 6 | 3 | 1 | 0

3. Primary Outcome: Number of Participants With Laboratory Test Abnormalities (Without Regard to Baseline Abnormality)
Description: Laboratory parameters included: hematology (hemoglobin, hematocrit, red blood cell, platelet and white blood cell count, neutrophils, eosinophils, monocytes, basophils and lymphocytes), chemistry (blood urea nitrogen, creatinine, sodium, potassium, aspartate aminotransferase, alanine aminotransferase, total bilirubin, alkaline phosphatase, albumin, total protein and serum pregnancy test [for all female participants]) and urine (urine pregnancy test [for all female participants]). Clinical significance of laboratory parameters was determined at the investigator's discretion.
Time Frame: Baseline up to 28 days after last dose of study treatment ( up to approximately 2 years)
Population: Population included all enrolled participants who received at least one dose of investigational product and with at least one observation of the given laboratory test during treatment period. Here, "number analyzed" signifies participant evaluable for each row.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1A: PF-06952229 20mg Monotherapy | Part 1A: PF-06952229 40mg Monotherapy | Part 1A: PF-06952229 80mg Monotherapy | Part 1A: PF-06952229 150mg Monotherapy | Part 1A: PF-06952229 250mg Monotherapy | Part 1A: PF-06952229 375mg Monotherapy | Part 1A: PF-06952229 500mg Monotherapy | Part 1B: PF-06952229 250mg + Enzalutamide | Part 1B: PF-06952229 375mg + Enzalutamide
Number analyzed (Participants) | 1 | 1 | 1 | 5 | 12 | 17 | 4 | 4 | 3
Participants
  HEMATOLOGY: Hemoglobin (g/dL) < 0.8xlower limit of normal (LLN) | 1 | 1 | 1 | 2 | 6 | 13 | 2 | 3 | 2
  HEMATOLOGY: Lymphocytes (10^3/mm^3) < 0.8xLLN | 0 | 0 | 1 | 3 | 8 | 9 | 2 | 2 | 1
  HEMATOLOGY: Basophils (10^3/mm^3) > 1.2xupper limit of normal (ULN) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
  HEMATOLOGY: Monocytes (10^3/mm^3) > 1.2xULN | 1 | 0 | 0 | 4 | 2 | 4 | 1 | 1 | 0
  HEMATOLOGY: Activated Partial Thromboplastin Time (sec) > 1.1xULN: number analyzed (Participants) | 1 | 1 | 1 | 5 | 9 | 17 | 4 | 4 | 3
  HEMATOLOGY: Activated Partial Thromboplastin Time (sec) > 1.1xULN | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 3 | 1
  HEMATOLOGY: Prothrombin Time (sec) > 1.1xULN: number analyzed (Participants) | 1 | 1 | 1 | 5 | 9 | 17 | 4 | 4 | 3
  HEMATOLOGY: Prothrombin Time (sec) > 1.1xULN | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
  HEMATOLOGY: Leukocytes (10^3/mm^3) < 0.6xLLN | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  HEMATOLOGY: Leukocytes (10^3/mm^3) > 1.5xULN | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  HEMATOLOGY: Neutrophils (10^3/mm^3) < 0.8xLLN | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  HEMATOLOGY: Neutrophils (10^3/mm^3)> 1.2xULN | 0 | 0 | 0 | 3 | 2 | 1 | 0 | 0 | 0
  HEMATOLOGY: Eosinophils (10^3/mm^3)> 1.2xULN | 1 | 1 | 0 | 1 | 2 | 7 | 3 | 0 | 2
  HEMATOLOGY: Prothrombin Intl. Normalized Ratio> 1.1xULN: number analyzed (Participants) | 1 | 1 | 1 | 5 | 9 | 17 | 4 | 4 | 3
  HEMATOLOGY: Prothrombin Intl. Normalized Ratio> 1.1xULN | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
  CLINICAL CHEMISTRY: Alkaline Phosphatase (U/L) > 3.0xULN: number analyzed (Participants) | 1 | 1 | 1 | 5 | 11 | 17 | 4 | 4 | 3
  CLINICAL CHEMISTRY: Alkaline Phosphatase (U/L) > 3.0xULN | 0 | 0 | 1 | 0 | 3 | 2 | 0 | 0 | 0
  CLINICAL CHEMISTRY: Urate (mg/dL) > 1.2xULN: number analyzed (Participants) | 1 | 1 | 1 | 5 | 9 | 17 | 4 | 4 | 3
  CLINICAL CHEMISTRY: Urate (mg/dL) > 1.2xULN | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  CLINICAL CHEMISTRY: Sodium (mEq/L) < 0.95xLLN: number analyzed (Participants) | 1 | 1 | 1 | 5 | 11 | 17 | 4 | 4 | 3
  CLINICAL CHEMISTRY: Sodium (mEq/L) < 0.95xLLN | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  CLINICAL CHEMISTRY: Potassium (mEq/L) < 0.9xLLN: number analyzed (Participants) | 1 | 1 | 1 | 5 | 11 | 17 | 4 | 4 | 3
  CLINICAL CHEMISTRY: Potassium (mEq/L) < 0.9xLLN | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
  CLINICAL CHEMISTRY: Potassium (mEq/L) > 1.1xULN: number analyzed (Participants) | 1 | 1 | 1 | 5 | 11 | 17 | 4 | 4 | 3
  CLINICAL CHEMISTRY: Potassium (mEq/L) > 1.1xULN | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
  CLINICAL CHEMISTRY: Chloride (mEq/L)< 0.9xLLN: number analyzed (Participants) | 1 | 1 | 1 | 5 | 11 | 17 | 4 | 4 | 3
  CLINICAL CHEMISTRY: Chloride (mEq/L)< 0.9xLLN | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  CLINICAL CHEMISTRY: Magnesium (mg/dL)< 0.9xLLN: number analyzed (Participants) | 1 | 1 | 1 | 5 | 11 | 17 | 4 | 4 | 3
  CLINICAL CHEMISTRY: Magnesium (mg/dL)< 0.9xLLN | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 0
  CLINICAL CHEMISTRY: Phosphate (mg/dL)< 0.8xLLN: number analyzed (Participants) | 1 | 1 | 1 | 5 | 11 | 17 | 4 | 4 | 3
  CLINICAL CHEMISTRY: Phosphate (mg/dL)< 0.8xLLN | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 2 | 1
  CLINICAL CHEMISTRY: Phosphate (mg/dL)> 1.2xULN: number analyzed (Participants) | 1 | 1 | 1 | 5 | 11 | 17 | 4 | 4 | 3
  CLINICAL CHEMISTRY: Phosphate (mg/dL)> 1.2xULN | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0
  CLINICAL CHEMISTRY: Glucose (mg/dL)> 1.5xULN: number analyzed (Participants) | 1 | 1 | 1 | 5 | 11 | 17 | 4 | 4 | 3
  CLINICAL CHEMISTRY: Glucose (mg/dL)> 1.5xULN | 0 | 0 | 0 | 1 | 1 | 2 | 1 | 1 | 0
  CLINICAL CHEMISTRY: Bilirubin (mg/dL)> 1.5xULN: number analyzed (Participants) | 1 | 1 | 1 | 5 | 11 | 17 | 4 | 4 | 3
  CLINICAL CHEMISTRY: Bilirubin (mg/dL)> 1.5xULN | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  CLINICAL CHEMISTRY: Aspartate Aminotransferase (U/L)> 3.0xULN: number analyzed (Participants) | 1 | 1 | 1 | 5 | 11 | 17 | 4 | 4 | 3
  CLINICAL CHEMISTRY: Aspartate Aminotransferase (U/L)> 3.0xULN | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 1 | 0
  CLINICAL CHEMISTRY: Alanine Aminotransferase (U/L)> 3.0xULN: number analyzed (Participants) | 1 | 1 | 1 | 5 | 11 | 17 | 4 | 4 | 3
  CLINICAL CHEMISTRY: Alanine Aminotransferase (U/L)> 3.0xULN | 0 | 0 | 0 | 0 | 1 | 4 | 3 | 1 | 0
  CLINICAL CHEMISTRY: Urea Nitrogen (mg/dL)> 1.3xULN: number analyzed (Participants) | 1 | 1 | 1 | 5 | 11 | 17 | 4 | 4 | 3
  CLINICAL CHEMISTRY: Urea Nitrogen (mg/dL)> 1.3xULN | 0 | 0 | 0 | 2 | 1 | 2 | 0 | 0 | 0
  CLINICAL CHEMISTRY: Creatinine (mg/dL)> 1.3xULN: number analyzed (Participants) | 1 | 1 | 1 | 5 | 11 | 17 | 4 | 4 | 3
  CLINICAL CHEMISTRY: Creatinine (mg/dL)> 1.3xULN | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0
  URINALYSIS: URINE Protein (Scalar)≥ 1: number analyzed (Participants) | 1 | 0 | 1 | 4 | 10 | 17 | 4 | 4 | 3
  URINALYSIS: URINE Protein (Scalar)≥ 1 | 0 | 0 | 0 | 0 | 3 | 3 | 2 | 0 | 1
  URINALYSIS: URINE Hemoglobin (Scalar)≥ 1: number analyzed (Participants) | 1 | 0 | 1 | 4 | 9 | 17 | 4 | 4 | 3
  URINALYSIS: URINE Hemoglobin (Scalar)≥ 1 | 0 | 0 | 0 | 0 | 4 | 8 | 2 | 4 | 3

4. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of PF-06952229 (Part 1A)
Description: Cmax was directly observed from data. Cmax was defined as maximum observed plasma concentration.
Time Frame: 0 (pre dose), 0.5, 1, 2, 4, 6 and 12 hours (post dose) on Day 1 and 7 of cycle 1, 0 (pre dose), 0.5, 1, 2, 4, 6 and 12 hours (post dose) on Day 1 of cycle 2.
Population: Participants with advanced/metastatic tumors in PF-06952229 single agent dose escalation phase, who had sufficient information to estimate at least 1 of the pharmacokinetic (PK) parameters of interest. Here, "number analyzed" signifies participant evaluable for each row.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms/milliliter (ng/mL)
Arm/Group | Part 1A: PF-06952229 20mg Monotherapy | Part 1A: PF-06952229 40mg Monotherapy | Part 1A: PF-06952229 80mg Monotherapy | Part 1A: PF-06952229 150mg Monotherapy | Part 1A: PF-06952229 250mg Monotherapy | Part 1A: PF-06952229 375mg Monotherapy | Part 1A: PF-06952229 500mg Monotherapy
Number analyzed (Participants) | 1 | 1 | 1 | 5 | 13 | 17 | 4
nanograms/milliliter (ng/mL)
  Cycle 1 Day 1 | 203.0 | 215.0 | 345.0 | 509.7 (173) | 1148 (65) | 1782 (117) | 1309 (309)
  Cycle 1 Day 7: number analyzed (Participants) | 1 | 1 | 1 | 4 | 6 | 15 | 4
  Cycle 1 Day 7 | 222.0 | 255.0 | 618.0 | 1050 (85) | 1787 (131) | 2727 (98) | 2917 (88)
  Cycle 2 Day 1: number analyzed (Participants) | 1 | 1 | 1 | 4 | 6 | 12 | 4
  Cycle 2 Day 1 | 128.0 | 240.0 | 200.0 | 696.0 (112) | 1019 (158) | 1876 (95) | 2434 (137)

5. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of PF-06952229 (Part 1B)
Description: Cmax was directly observed from data. Cmax was defined as maximum observed plasma concentration.
Time Frame: 0 (pre dose), 0.5, 1, 2, 4, 6 and 12 hours (post dose) on Day 1 and 21 of cycle 1, 0 (pre dose), 0.5, 1, 2, 4, 6 and 12 hours (post dose) on Day 1 of cycle 2.
Population: Participants with metastatic castration-resistant prostate cancer (mCRPC), conducted dose escalation of PF-06952229 in combination with enzalutamide, who had sufficient information to estimate at least 1 of the PK parameters of interest. Here, "number analyzed" signifies participant evaluable for each row
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part 1B: PF-06952229 250mg + Enzalutamide | Part 1B: PF-06952229 375mg + Enzalutamide
Number analyzed (Participants) | 4 | 3
ng/mL
  Cycle 1 Day 1 | 1619 (45) | 1462 (21)
  Cycle 1 Day 21: number analyzed (Participants) | 3 | 3
  Cycle 1 Day 21 | 1289 (35) | 1500 (32)
  Cycle 2 Day 1: number analyzed (Participants) | 3 | 3
  Cycle 2 Day 1 | 693.5 (84) | 960.3 (13)

6. Secondary Outcome: Time of Observed Maximum Plasma Concentration (Tmax) of PF-06952229 (Part 1A)
Description: Tmax was defined as time to maximum observed concentration. Observed directly from data as time of first occurrence.
Time Frame: as for outcome 4
Population: Participants with advanced/metastatic tumors in PF-06952229 single agent dose escalation phase, who had sufficient information to estimate at least 1 of the PK parameters of interest. Here, "number analyzed" signifies participant evaluable for each row.
Measure: Median (Full Range); unit: hour (hr)
Arm/Group | Part 1A: PF-06952229 20mg Monotherapy | Part 1A: PF-06952229 40mg Monotherapy | Part 1A: PF-06952229 80mg Monotherapy | Part 1A: PF-06952229 150mg Monotherapy | Part 1A: PF-06952229 250mg Monotherapy | Part 1A: PF-06952229 375mg Monotherapy | Part 1A: PF-06952229 500mg Monotherapy
Number analyzed (Participants) | 1 | 1 | 1 | 5 | 13 | 17 | 4
hour (hr)
  Cycle 1 Day 1 | 2.10 [2.10 to 2.10] | 3.83 [3.83 to 3.83] | 2.00 [2.00 to 2.00] | 2.15 [1.08 to 5.83] | 2.17 [1.00 to 9.00] | 2.03 [0.950 to 9.00] | 1.97 [1.00 to 2.12]
  Cycle 1 Day 7: number analyzed (Participants) | 1 | 1 | 1 | 4 | 6 | 15 | 4
  Cycle 1 Day 7 | 0.967 [0.967 to 0.967] | 2.05 [2.05 to 2.05] | 2.18 [2.18 to 2.18] | 1.51 [0.450 to 2.38] | 2.00 [0 to 3.90] | 1.92 [0.850 to 4.33] | 1.48 [1.00 to 2.00]
  Cycle 2 Day 1: number analyzed (Participants) | 1 | 1 | 1 | 4 | 6 | 12 | 4
  Cycle 2 Day 1 | 3.95 [3.95 to 3.95] | 6.08 [6.08 to 6.08] | 5.52 [5.52 to 5.52] | 5.99 [1.00 to 6.03] | 4.14 [1.03 to 5.93] | 5.02 [1.00 to 9.08] | 3.65 [2.00 to 9.00]

7. Secondary Outcome: Time of Observed Maximum Plasma Concentration (Tmax) of PF-06952229 (Part 1B)
Description: Tmax was defined as time to maximum observed concentration. Observed directly from data as time of first occurrence.
Time Frame: as for outcome 5
Population: Participants with mCRPC, conducted dose escalation of PF-06952229 in combination with enzalutamide, who had sufficient information to estimate at least 1 of the PK parameters of interest. Here, "number analyzed" signifies participant evaluable for each row.
Measure: Median (Full Range); unit: hour (hr)
Arm/Group | Part 1B: PF-06952229 250mg + Enzalutamide | Part 1B: PF-06952229 375mg + Enzalutamide
Number analyzed (Participants) | 4 | 3
hour (hr)
  Cycle 1 Day 1 | 2.20 [2.03 to 5.73] | 1.98 [1.95 to 2.00]
  Cycle 1 Day 21: number analyzed (Participants) | 3 | 3
  Cycle 1 Day 21 | 1.00 [0.967 to 2.20] | 0.983 [0.917 to 1.85]
  Cycle 2 Day 1: number analyzed (Participants) | 3 | 3
  Cycle 2 Day 1 | 2.05 [1.83 to 3.68] | 2.00 [1.95 to 2.00]

8. Secondary Outcome: Area Under the Plasma Concentration-Time Profile From Time Zero to Time of the Last Quantifiable Concentration (AUClast) of PF-06952229 (Part 1A)
Description: AUClast was area under the plasma concentration time-curve from zero (pre-dose) to the last measured concentration.
Time Frame: 0 (pre dose), 0.5, 1, 2, 4, 6 and 12 hours (post dose) on Day 1 of cycle 1 and cycle 2
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms*hour/milliliter (ng*hr/mL)
Arm/Group | Part 1A: PF-06952229 20mg Monotherapy | Part 1A: PF-06952229 40mg Monotherapy | Part 1A: PF-06952229 80mg Monotherapy | Part 1A: PF-06952229 150mg Monotherapy | Part 1A: PF-06952229 250mg Monotherapy | Part 1A: PF-06952229 375mg Monotherapy | Part 1A: PF-06952229 500mg Monotherapy
Number analyzed (Participants) | 1 | 1 | 1 | 5 | 13 | 17 | 4
nanograms*hour/milliliter (ng*hr/mL)
  Cycle 1 Day 1 | 785.0 | 1010 | 1190 | 2726 (136) | 5111 (72) | 8470 (133) | 6401 (281)
  Cycle 2 Day 1: number analyzed (Participants) | 1 | 1 | 1 | 4 | 6 | 12 | 4
  Cycle 2 Day 1 | 466.0 | 547.0 | 508.0 | 2035 (42) | 3130 (329) | 10050 (97) | 10540 (159)

9. Secondary Outcome: Area Under the Plasma Concentration-Time Profile From Time Zero to Time of the Last Quantifiable Concentration (AUClast) of PF-06952229 (Part 1B)
Description: AUClast was area under the plasma concentration time-curve from zero (pre-dose) to the last measured concentration.
Time Frame: 0 (pre dose), 0.5, 1, 2, 4, 6 and 12 hours (post dose) on Day 1 of cycle 1 and cycle 2
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Part 1B: PF-06952229 250mg + Enzalutamide | Part 1B: PF-06952229 375mg + Enzalutamide
Number analyzed (Participants) | 4 | 3
ng*hr/mL
  Cycle 1 Day 1 | 16940 (24) | 13430 (34)
  Cycle 2 Day 1: number analyzed (Participants) | 3 | 3
  Cycle 2 Day 1 | 6707 (85) | 5656 (11)

10. Secondary Outcome: Area Under the Plasma Concentration-Time Profile From Time Zero Extrapolated to Infinite Time (AUCinf) of PF-06952229 (Part 1A)
Description: AUCinf was defined as area under the plasma concentration-time curve from time zero to infinity.
Time Frame: 0 (pre dose), 0.5, 1, 2, 4, 6 and 12 hours (post dose) on Day 1 of cycle 1 and cycle 2
Population: Participants with advanced/metastatic tumors in PF-06952229 single agent dose escalation phase, who had sufficient information to estimate at least 1 of the PK parameters of interest and contributed to the summary statistics for AUCinf. AUCinf can be evaluated only when a well characterized terminal phase was observed, which is defined as one with at least 3 data points, r^2≥0.9, and AUCextrap%≤20. Here, "number analyzed" signifies participant evaluable for each row.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Part 1A: PF-06952229 20mg Monotherapy | Part 1A: PF-06952229 40mg Monotherapy | Part 1A: PF-06952229 80mg Monotherapy | Part 1A: PF-06952229 150mg Monotherapy | Part 1A: PF-06952229 250mg Monotherapy | Part 1A: PF-06952229 375mg Monotherapy | Part 1A: PF-06952229 500mg Monotherapy
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 2 | 1
ng*hr/mL
  Cycle 1 Day 1 |  |  |  |  | 4974 (32) | 10160 (43) | 18500
  Cycle 2 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Cycle 2 Day 1 |  |  |  |  |  | 6820 |

11. Secondary Outcome: Area Under the Plasma Concentration-Time Profile From Time Zero Extrapolated to Infinite Time (AUCinf) of PF-06952229 (Part 1B)
Description: AUCinf was defined as area under the plasma concentration-time curve from time zero to infinity.
Time Frame: 0 (pre dose), 0.5, 1, 2, 4, 6 and 12 hours (post dose) on Day 1 of cycle 1 and cycle 2
Population: Participants with mCRPC, conducted dose escalation of PF-06952229 in combination with enzalutamide, who had sufficient information to estimate at least 1 of the PK parameters of interest and contributed to the summary statistics for AUCinf. AUCinf can be evaluated only when a well characterized terminal phase was observed, which is defined as one with at least 3 data points, r^2≥0.9, and AUCextrap%≤20. Here, "number analyzed" signifies participant evaluable for each row.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Part 1B: PF-06952229 250mg + Enzalutamide | Part 1B: PF-06952229 375mg + Enzalutamide
Number analyzed (Participants) | 2 | 2
ng*hr/mL
  Cycle 1 Day 1 | 17100 (1) | 14750 (61)
  Cycle 2 Day 1 | 5095 (75) | 6214 (3)

12. Secondary Outcome: Apparent Clearance (CL/F) of PF-06952229 (Part 1A)
Description: Apparent Clearance After Oral Dose (CL/F) was defined as apparent clearance after oral dose on the last day of treatment period. CL/F = Dose/AUCinf for single dose; CL/F = Dose/AUCtau for steady-state. AUCtau was defined as Area under the plasma concentration-time profile from time zero to time tau (τ), the dosing interval, where τ = 24 and 12 hours for QD and BID dosing, respectively.
Time Frame: as for outcome 4
Population: Participants with advanced/metastatic tumors in PF-06952229 single agent dose escalation phase, who had sufficient information to estimate at least 1 of the PK parameters of interest and contributed to the summary statistics for CL/F. CL/F can be evaluated only when a well characterized terminal phase was observed, which is defined as one with at least 3 data points, r^2≥0.9, and AUCextrap%≤20. Here, "number analyzed" signifies participant evaluable for each row.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter per hour (L/hr)
Arm/Group | Part 1A: PF-06952229 20mg Monotherapy | Part 1A: PF-06952229 40mg Monotherapy | Part 1A: PF-06952229 80mg Monotherapy | Part 1A: PF-06952229 150mg Monotherapy | Part 1A: PF-06952229 250mg Monotherapy | Part 1A: PF-06952229 375mg Monotherapy | Part 1A: PF-06952229 500mg Monotherapy
Number analyzed (Participants) | 1 | 1 | 1 | 4 | 6 | 15 | 4
liter per hour (L/hr)
  Cycle 1 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 2 | 1
  Cycle 1 Day 1 |  |  |  |  | 50.23 (32) | 36.86 (43) | 27.10
  Cycle 1 Day 7 | 9.850 | 21.80 | 22.30 | 17.36 (79) | 15.95 (127) | 19.49 (92) | 29.04 (132)
  Cycle 2 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Cycle 2 Day 1 |  |  |  |  |  | 55.00 |

13. Secondary Outcome: Apparent Clearance (CL/F) of PF-06952229 (Part 1B)
Description: as for outcome 12
Time Frame: as for outcome 5
Population: Participants with mCRPC, conducted dose escalation of PF-06952229 in combination with enzalutamide, who had sufficient information to estimate at least 1 of the PK parameters of interest and contributed to the summary statistics for CL/F. CL/F can be evaluated only when a well characterized terminal phase was observed, which is defined as one with at least 3 data points, r^2≥0.9, and AUCextrap%≤20. Here, "number analyzed" signifies participant evaluable for each row.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/hr
Arm/Group | Part 1B: PF-06952229 250mg + Enzalutamide | Part 1B: PF-06952229 375mg + Enzalutamide
Number analyzed (Participants) | 3 | 3
L/hr
  Cycle 1 Day 1: number analyzed (Participants) | 2 | 2
  Cycle 1 Day 1 | 14.65 (0) | 25.38 (62)
  Cycle 1 Day 21 | 30.86 (26) | 43.04 (41)
  Cycle 2 Day 1: number analyzed (Participants) | 2 | 2
  Cycle 2 Day 1 | 49.06 (76) | 60.39 (3)

14. Secondary Outcome: Apparent Volume of Distribution (Vz/F) of PF-06952229 (Part 1A)
Description: Vz/F was defined as apparent volume of distribution. Vz/F = Dose / (AUCinf* kel) for single dose; Vz/F = Dose / (AUCtau* kel) for steady-state. AUCtau was defined as Area under the plasma concentration-time profile from time zero to time tau (τ), the dosing interval, where τ = 24 and 12 hours for QD and BID dosing, respectively. Kel was defined as terminal phase rate constant.
Time Frame: as for outcome 4
Population: Participants with advanced/metastatic tumors in PF-06952229 single agent dose escalation phase, who had sufficient information to estimate at least 1 of the PK parameters of interest and contributed to the summary statistics for Vz/F. Vz/F can be evaluated only when a well characterized terminal phase was observed, which is defined as one with at least 3 data points, r^2≥0.9, and AUCextrap%≤20. Here, "number analyzed" signifies participant evaluable for each row.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter (L)
Arm/Group | Part 1A: PF-06952229 20mg Monotherapy | Part 1A: PF-06952229 40mg Monotherapy | Part 1A: PF-06952229 80mg Monotherapy | Part 1A: PF-06952229 150mg Monotherapy | Part 1A: PF-06952229 250mg Monotherapy | Part 1A: PF-06952229 375mg Monotherapy | Part 1A: PF-06952229 500mg Monotherapy
Number analyzed (Participants) | 0 | 1 | 0 | 0 | 2 | 2 | 1
liter (L)
  Cycle 1 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 2 | 1
  Cycle 1 Day 1 |  |  |  |  | 187.2 (31) | 178.1 (46) | 130.0
  Cycle 1 Day 7: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 1 | 1
  Cycle 1 Day 7 |  | 139.0 |  |  |  | 287.0 | 665.0
  Cycle 2 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Cycle 2 Day 1 |  |  |  |  |  | 266.0 |

15. Secondary Outcome: Apparent Volume of Distribution (Vz/F) of PF-06952229 (Part 1B)
Description: as for outcome 14
Time Frame: 0 (pre dose), 0.5, 1, 2, 4, 6 and 12 hours (post dose) on Day 1 of cycle 1 and cycle 2
Population: Participants with mCRPC, conducted dose escalation of PF-06952229 in combination with enzalutamide, who had sufficient information to estimate at least 1 of the PK parameters of interest and contributed to the summary statistics for Vz/F. Vz/F can be evaluated only when a well characterized terminal phase was observed, which is defined as one with at least 3 data points, r^2≥0.9, and AUCextrap%≤20. Here, "number analyzed" signifies participant evaluable for each row.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter
Arm/Group | Part 1B: PF-06952229 250mg + Enzalutamide | Part 1B: PF-06952229 375mg + Enzalutamide
Number analyzed (Participants) | 2 | 2
Liter
  Cycle 1 Day 1 | 161.8 (14) | 228.4 (4)
  Cycle 2 Day 1 | 372.4 (67) | 408.7 (11)

16. Secondary Outcome: Terminal Elimination Half-Life (T1/2) of PF-06952229 (Part 1A)
Description: Plasma terminal elimination half-life (T1/2) was the time measured for the plasma concentration to decrease by one half of its initial concentration.
Time Frame: as for outcome 4
Population: Participants with advanced/metastatic tumors in PF-06952229 single agent dose escalation phase, who had sufficient information to estimate at least 1 of the PK parameters of interest and contributed to the summary statistics for T1/2. T1/2 can be evaluated only when a well characterized terminal phase was observed, which is defined as one with at least 3 data points, r^2≥0.9, and AUCextrap%≤20. Here, "number analyzed" signifies participant evaluable for each row.
Measure: Mean (Standard Deviation); unit: Hour
Arm/Group | Part 1A: PF-06952229 20mg Monotherapy | Part 1A: PF-06952229 40mg Monotherapy | Part 1A: PF-06952229 80mg Monotherapy | Part 1A: PF-06952229 150mg Monotherapy | Part 1A: PF-06952229 250mg Monotherapy | Part 1A: PF-06952229 375mg Monotherapy | Part 1A: PF-06952229 500mg Monotherapy
Number analyzed (Participants) | 0 | 1 | 0 | 0 | 2 | 2 | 1
Hour
  Cycle 1 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 2 | 1
  Cycle 1 Day 1 |  |  |  |  | 2.585 (0.021213) | 3.345 (0.077782) | 3.320
  Cycle 1 Day 7: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 1 | 1
  Cycle 1 Day 7 |  | 4.410 |  |  |  | 2.550 | 3.670
  Cycle 2 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Cycle 2 Day 1 |  |  |  |  |  | 3.350 |

17. Secondary Outcome: Terminal Elimination Half-Life (T1/2) of PF-06952229 (Part 1B)
Description: as for outcome 16
Time Frame: 0 (pre dose), 0.5, 1, 2, 4, 6 and 12 hours (post dose) on Day 1 of cycle 1 and cycle 2
Population: Participants with mCRPC, conducted dose escalation of PF-06952229 in combination with enzalutamide, who had sufficient information to estimate at least 1 of the PK parameters of interest and contributed to the summary statistics for T1/2. T1/2 can be evaluated only when a well characterized terminal phase was observed, which is defined as one with at least 3 data points, r^2≥0.9, and AUCextrap%≤20. Here, "number analyzed" signifies participant evaluable for each row.
Measure: Mean (Standard Deviation); unit: Hour
Arm/Group | Part 1B: PF-06952229 250mg + Enzalutamide | Part 1B: PF-06952229 375mg + Enzalutamide
Number analyzed (Participants) | 2 | 2
Hour
  Cycle 1 Day 1 | 7.700 (1.0041) | 6.670 (3.3658)
  Cycle 2 Day 1 | 5.265 (0.33234) | 4.700 (0.39598)

18. Secondary Outcome: Number of Participants With Prostate Specific Antigen 50 (PSA50) Response
Description: Prostate-specific antigen decline by more than 50% from baseline was analyzed. PSA partial response was defined as a ≥50% decline in PSA from Cycle 1 Day 1 (baseline) PSA value. This PSA decline much be confirmed to be sustained by a second PSA value obtained 4 or more weeks later.
Time Frame: Baseline, Cycle 1 Day 1 (at the beginning of Cycle 1), and then every 3 cycles (each cycle is 28 days) until end of treatment (an average of 1 year)
Population: Population included all enrolled participants who had metastatic castration resistant prostate cancer (mCRPC)
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1A: PF-06952229 20mg Monotherapy | Part 1A: PF-06952229 40mg Monotherapy | Part 1A: PF-06952229 80mg Monotherapy | Part 1A: PF-06952229 150mg Monotherapy | Part 1A: PF-06952229 250mg Monotherapy | Part 1A: PF-06952229 375mg Monotherapy | Part 1A: PF-06952229 500mg Monotherapy | Part 1B: PF-06952229 250mg + Enzalutamide | Part 1B: PF-06952229 375mg + Enzalutamide
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 8 | 14 | 4 | 4 | 3
Participants | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0

19. Secondary Outcome: Percentage of Participants With Objective Response
Description: Percentage of participants with objective response based assessment of confirmed complete response (CR) or confirmed partial response (PR). Complete response was defined as complete disappearance of all target lesions with the exception of nodal disease. All target nodes must decrease to normal size (short axis <10 mm). All target lesions must be assessed. Partial response was defined as greater than or equal to 30% decrease under baseline of the sum of diameters of all target measurable lesions. The short diameter was used in the sum for target nodes, while the longest diameter was used in the sum for all other target lesions. All target lesions must be assessed.
Time Frame: Baseline and every 8 to 12 weeks through time of confirmed disease progression, unacceptable toxicity, or through study completion, approximately 2 years.
Population: Population included all enrolled participants who received at least 1 dose of investigational product, had baseline assessment and at least 1 post baseline assessment, disease progression, or death before the first tumor assessment.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Part 1A: PF-06952229 20mg Monotherapy | Part 1A: PF-06952229 40mg Monotherapy | Part 1A: PF-06952229 80mg Monotherapy | Part 1A: PF-06952229 150mg Monotherapy | Part 1A: PF-06952229 250mg Monotherapy | Part 1A: PF-06952229 375mg Monotherapy | Part 1A: PF-06952229 500mg Monotherapy | Part 1B: PF-06952229 250mg + Enzalutamide | Part 1B: PF-06952229 375mg + Enzalutamide
Number analyzed (Participants) | 1 | 1 | 1 | 5 | 10 | 14 | 4 | 4 | 2
Percentage of participants | 0 [0.0 to 97.5] | 0 [0.0 to 97.5] | 0 [0.0 to 97.5] | 0 [0.0 to 52.2] | 0 [0.0 to 30.8] | 7.1 [0.2 to 33.9] | 0 [0.0 to 60.2] | 0 [0.0 to 60.2] | 0 [0.0 to 84.2]

ADVERSE EVENTS:
Time Frame: Baseline up to 28 days after last dose of study treatment ( up to approximately 2 years)
Description: The same event may appear as both an adverse event (AE) and an serious adverse event (SAE). An event may be categorized as serious in one participant and as non-serious in another participant, or one participant may have experienced both a serious and non-serious event during the study. Total number at risk below refers to the number of participants evaluable for SAEs or AEs.
Arm/Group | Part 1A: PF-06952229 20mg Monotherapy | Part 1A: PF-06952229 40mg Monotherapy | Part 1A: PF-06952229 80mg Monotherapy | Part 1A: PF-06952229 150mg Monotherapy | Part 1A: PF-06952229 250mg Monotherapy | Part 1A: PF-06952229 375mg Monotherapy | Part 1A: PF-06952229 500mg Monotherapy | Part 1B: PF-06952229 250mg + Enzalutamide | Part 1B: PF-06952229 375mg + Enzalutamide
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/1 | 0/1 | 1/5 | 0/13 | 0/17 | 0/4 | 0/4 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1 | 0/1 | 3/5 | 3/13 | 5/17 | 0/4 | 0/4 | 0/3
Other Adverse Events (participants affected / at risk) | 1/1 | 1/1 | 1/1 | 4/5 | 13/13 | 16/17 | 4/4 | 4/4 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1A: PF-06952229 20mg Monotherapy (N=1) | Part 1A: PF-06952229 40mg Monotherapy (N=1) | Part 1A: PF-06952229 80mg Monotherapy (N=1) | Part 1A: PF-06952229 150mg Monotherapy (N=5) | Part 1A: PF-06952229 250mg Monotherapy (N=13) | Part 1A: PF-06952229 375mg Monotherapy (N=17) | Part 1A: PF-06952229 500mg Monotherapy (N=4) | Part 1B: PF-06952229 250mg + Enzalutamide (N=4) | Part 1B: PF-06952229 375mg + Enzalutamide (N=3)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Mouth haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Disease progression (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hepatic haemorrhage (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Intracranial tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Laryngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1A: PF-06952229 20mg Monotherapy (N=1) | Part 1A: PF-06952229 40mg Monotherapy (N=1) | Part 1A: PF-06952229 80mg Monotherapy (N=1) | Part 1A: PF-06952229 150mg Monotherapy (N=5) | Part 1A: PF-06952229 250mg Monotherapy (N=13) | Part 1A: PF-06952229 375mg Monotherapy (N=17) | Part 1A: PF-06952229 500mg Monotherapy (N=4) | Part 1B: PF-06952229 250mg + Enzalutamide (N=4) | Part 1B: PF-06952229 375mg + Enzalutamide (N=3)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 1 | 1 | 1 | 6 | 1 | 1 | 1
Eosinophilia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lymph node pain (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Atrial flutter (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Adrenal insufficiency (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Ocular hyperaemia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Visual impairment (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 2 | 0 | 1 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 1 | 2 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Gingival bleeding (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Mouth haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 1 | 2 | 5 | 4 | 3 | 1 | 0
Proctalgia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 6 | 1 | 2 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Chills (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 1 | 0 | 0 | 1 | 1 | 4 | 2 | 0 | 0
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Mucosal inflammation (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0
Temperature intolerance (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cystitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Osteomyelitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 2 | 7 | 3 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 2 | 7 | 3 | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Brain natriuretic peptide increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
International normalised ratio increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Prostatic specific antigen increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
SARS-CoV-2 test positive (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Troponin I increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 1 | 2 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 3 | 1 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 2 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1 | 2 | 0 | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1 | 2 | 0 | 0 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 2 | 3 | 5 | 3 | 2 | 0
Hemiparesis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0
Bladder spasm (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 1
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0
Urinary tract pain (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 3 | 2 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2 | 2 | 1 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 2 | 2 | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0

LIMITATIONS AND CAVEATS:
The trial began on 04 October 2018 with LPLV occurring on 30 March 2022 following Pfizer's strategic decision (not due to any specific safety reasons or request from a regulatory authority) to terminate the study, which included the period during which the COVID-19 pandemic was occurring globally since 11 March 2020.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2021-05-07): https://cdn.clinicaltrials.gov/large-docs/91/NCT03685591/Prot_000.pdf
  • Statistical Analysis Plan (2022-05-20): https://cdn.clinicaltrials.gov/large-docs/91/NCT03685591/SAP_001.pdf